CLINICAL TRIAL: NCT05674123
Title: Feasibility of Transanal Robot-Assisted Resection of Distal Colorectal Lesions Using the Medrobotics Flex® System: A Pilot Study
Brief Title: Evaluating the Safety and Effectiveness of the Flex Robotic System for the Surgical Removal of Colorectal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 19-009663; NCI-2022-09474 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-009663 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2022-12-12; First posted 2023-01-06 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Neoplasm
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy; Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Device Feasibility (Flex Robotic System) (Experimental): Patients undergo resection with Flex Robotic System on study. Patients also undergo colonoscopy with or without rectal endoscopic ultrasound at screening.
  Interventions: Procedure: Colonoscopy; Procedure: Endoscopic Ultrasound; Other: Medical Chart Review; Other: Medical Device Usage and Evaluation; Procedure: Resection

INTERVENTIONS:
Procedure: Colonoscopy — Undergo colonoscopy
Procedure: Endoscopic Ultrasound — Undergo rectal endoscopic ultrasound
  Other Names: endosonography; EUS
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review
Other: Medical Device Usage and Evaluation — Undergo resection with the Flex Robotic System
Procedure: Resection — Undergo resection with the Flex Robotic System
  Other Names: Robot-assisted surgical Resection

SUMMARY:
This clinical trial assesses the safety and effectiveness of a new device called the Flex Robotic System in the surgical removal (resection) of colorectal lesions. When an area of abnormal tissue called a lesion is found in the colon or rectum, it is often not known if the lesion is cancerous or non-cancerous. Recommendation to remove the lesion may be made. Current methods of resection can be challenging and time-consuming. The Flex Robotic System is a new device that provides a stable working environment, better ability to grasp and cut lesions, and better tissue handling when performing a resection. The Flex Robotic system may be more effective at removing colorectal lesions than standard resection techniques.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the rates of complete en bloc resection and adverse events of the Flex Robotic System for distal colorectal lesions.

OUTLINE:

Patients undergo resection with Flex Robotic System on study. Patients also undergo colonoscopy with or without rectal endoscopic ultrasound at screening.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 22 years (minimum age approved for use)
* Polypoid (0-Is) and non-polypoid (0-IIa, 0-IIb and 0-IIc) lateral spreading lesions according to Paris classification
* Colorectal lesions situated between 5 and 15 cm from the dentate line
* Colorectal mucosal lesions ranging from 1.5 to 7 cm in maximum diameter
* Colorectal subepithelial lesions < 2 cm in size
* Absence of uncorrectable bleeding disorder or coagulopathy
* Platelet count > 50,000
* International normalized ratio (INR) < 1.5
* Ability to give informed consent

Exclusion Criteria:

* Inability to receive general anesthesia
* Presence of medical conditions for which a transanal approach is contraindicated (e.g., anal stricture, radiation proctopathy)
* Excavated (0-III) colorectal lesions according to Paris classification
* Suboptimal colon preparation
* Clinical discretion of the provider

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Rates of complete en bloc resection | Up to 2 years
  Rates of complete en bloc resection
Incidence of adverse events | Up to 2 years
  The primary endpoint will be the Incidence of adverse events using the Flex Robotic System for distal colorectal lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Louis M Wong Kee Song, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States